CLINICAL TRIAL: NCT07286149
Title: KEYMAKER-U01 Substudy 01F: A Phase 1b/2 Umbrella Study With Rolling Arms of Investigational Agents for Previously Treated Participants With Advanced or Metastatic Nonsquamous Non-small Cell Lung Cancer (NSCLC) With KRAS G12C Mutations
Brief Title: A Clinical Study of MK-1084 With Other Treatments for Non-small Cell Lung Cancer (MK-3475-01F)
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 3475-01F; MK-3475-01F (Other: MSD); 2024-512248-47-00 (Registry Identifier: EU CT); U1111-1304-4707 (Registry Identifier: UTN)
Record Dates: First submitted 2025-11-17; First posted 2025-12-16 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Lung Neoplasm Malignant
MeSH Terms: conditions — Lung Neoplasms | interventions — patritumab deruxtecan; Cetuximab

STUDY DESIGN:
Intervention Model Description: Participants will be enrolled and treated sequentially during dose escalation followed by parallel assignment in the expansion phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MK-1084 + Patritumab deruxtecan (HER3-DXd) (Experimental): Participants will receive MK-1084 and HER3-DXd until discontinuation due to toxicity, adverse event (AE) or at the discretion of an investigator.
  Interventions: Drug: MK-1084; Biological: Patritumab deruxtecan
- MK-1084 + Sacituzumab tirumotecan (Sac-TMT) (Experimental): Participants will receive MK-1084 and sac-TMT until discontinuation due to toxicity, AE or at the discretion of an investigator.
  Interventions: Drug: MK-1084; Biological: Sacituzumab tirumotecan; Drug: Rescue Medications
- MK-1084 + Cetuximab (Experimental): Participants will receive MK-1084 and cetuximab until discontinuation due to toxicity, AE or at the discretion of an investigator.
  Interventions: Drug: MK-1084; Biological: Cetuximab

INTERVENTIONS:
Drug: MK-1084 — Oral administration
Biological: Patritumab deruxtecan — IV infusion
  Other Names: HER3-DXd; MK-1022; U3-1402
  Arms: MK-1084 + Patritumab deruxtecan (HER3-DXd)
Biological: Sacituzumab tirumotecan — IV Infusion
  Other Names: Sac-TMT; MK-2870; SKB264
  Arms: MK-1084 + Sacituzumab tirumotecan (Sac-TMT)
Biological: Cetuximab — IV Infusion
  Other Names: C225; Erbitux
  Arms: MK-1084 + Cetuximab
Drug: Rescue Medications — Participants receive rescue medication at the investigator's discretion, per approved product label. Recommended rescue medications are histamine -1 (H1) receptor agonist, histamine-2 (H2) receptor antagonist, acetaminophen or equivalent, dexamethasone or equivalent infusion, or steroid mouthwash (dexamethasone or equivalent) for prevention of chemotherapy induced nausea and vomiting.
  Arms: MK-1084 + Sacituzumab tirumotecan (Sac-TMT)

SUMMARY:
Researchers want to learn if MK-1084, the study medicine, can treat advanced or metastatic non-squamous NSCLC. MK-1084 is a targeted therapy, which is a treatment that works to control how specific types of cancer cells grow and spread. The goals of this study are to learn:

* About the safety of MK-1084 and if people tolerate it when taken with other treatments
* How many people have the cancer respond (get smaller or go away) to the treatments

DETAILED DESCRIPTION:
This is a substudy of the master protocol MK-3475-U01 (KEYMAKER-U01) - NCT04165798.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has histologically or cytologically confirmed diagnosis of advanced or metastatic non-squamous non-small cell lung cancer (NSCLC)
* Has tumor tissue or circulating tumor deoxyribonucleic acid (ctDNA) that demonstrates the presence of Kirsten rat sarcoma viral oncogene (KRAS) mutation of glycine to cysteine at codon 12 (G12C) mutations
* Has documented disease progression after receiving 1-2 prior lines of programmed cell death protein 1 (PD-1)/programmed death-ligand 1 (PD-L1) therapy and platinum-based chemotherapy
* Provides archival tumor tissue sample of a tumor lesion not previously irradiated
* Has provided tissue prior to treatment allocation/randomization from a newly obtained biopsy of a tumor lesion not previously irradiated
* Participants with human immunodeficiency virus (HIV) infection must have well-controlled HIV on antiretroviral therapy (ART) per protocol

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has a diagnosis of small cell lung cancer or, for mixed tumors, presence of small cell elements
* Has clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has active inflammatory bowel disease requiring immunosuppressive medication or previous history of inflammatory bowel disease
* Has evidence of any leptomeningeal disease
* Has uncontrolled or significant cardiovascular disorder or cerebrovascular disease prior to allocation/randomization
* Has one or more of the following ophthalmological conditions: a) Clinically significant corneal disease b) history of documented severe dry eye syndrome, severe Meibomian gland disease and/or blepharitis
* HIV-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease
* Has received previous treatment with an agent targeting KRAS
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study intervention
* Has known additional malignancy that is progressing or has required active treatment within the past 3 years
* Has history of (noninfectious) pneumonitis/ interstitial lung disease (ILD) that required steroids or has current pneumonitis/ILD
* Has an active infection requiring systemic therapy
* Have not adequately recovered from major surgery or have ongoing surgical complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2026-02-23 (Estimated); Primary Completion 2031-08-11 (Estimated); Study Completion 2036-07-20 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experience a Dose Limiting Toxicity (DLT) | Up to 42 days
  DLT will be defined as any drug-related AE observed during the DLT evaluation period (up to 42 days) that results in a change to a given dose or a delay in initiating the next treatment.
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 65 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants that experience AEs will be reported.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 64 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants that discontinue study intervention due to an AE will be reported.
Objective Response Rate (ORR) | Up to approximately 65 months
  ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1). The percentage of participants who experience CR or PR as assessed by Blinded Independent Central Review (BICR) will be presented.

SECONDARY OUTCOMES:
Duration of Response (DOR) | Up to approximately 65 months
  For participants who demonstrate a confirmed CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR as assessed by BICR will be presented.
Progression-Free Survival (PFS) | Up to approximately 124 months
  PFS is defined as the time from randomization to the first documented PD or death due to any cause, whichever occurs first as assessed by RECIST 1.1. PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by BICR will be presented.
Area Under the Curve From Time 0 to the End of the Dosing Interval (AUC tau) | Predose and at designated time points post-dose (up to approximately 65 months)
  Blood samples will be collected at multiple time points to estimate AUC tau.
Maximum Plasma Concentration (Cmax) | Predose and at designated time points post-dose (up to approximately 65 months)
  Blood samples will be collected at multiple time points to estimate Cmax.
Minimum Observed Concentration (Ctrough) | Predose and at designated time points post-dose (up to approximately 65 months)
  Blood samples will be collected at multiple time points to estimate Ctrough.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com